CLINICAL TRIAL: NCT01776502
Title: A Prospective, Non Randomized, Open, Multicenter Trial to Evaluate Non Specific Symptoms and Quality of Life (SF 36) Before and After Surgery for Mild Primary Hyperparathyroidism
Brief Title: Evaluation of Non Specific Symptoms and Quality of Life Before and After Surgery for Mild Primary Hyperparathyroidism
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0255
Record Dates: First submitted 2012-10-24; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Primary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Hyperparathyroidism: The cohort of patients is made of patients with primary mild hyperparathyroidism and who have received a surgery at Nantes, Angers, Limoges or Marseille University Hospitals

SUMMARY:
The purpose of this study is to evaluate the evolution of the non specific symptoms for 116 patients with mild primary hyperparathyroidism before and 3, 6 and 12 months after surgery. A clinical score predicting clinical improvement at one year will be created.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with known moderate HPTI will be considered for participation.

Patients with sporadic mild HPTI defined by:

* calcemia > 2.6 mmol/L , PTH > 25 ng/L and creatininemia < 160µmol/L OR
* calcemia between 2.5 and 2.6 mmol/L and PTH > 35 ng/L
* calcemia ≤2.85 mmol/L
* urine calcium level / 24 hours < 10 mmol (400 mg),
* decrease of the creatinin's clearance : 30% lower than normal population with the same age
* patients younger than 50
* patients who can't be followed

Exclusion Criteria:

* familial hypercalcemia
* multiple endocrinal neoplasia
* treatment with lithium or thiazides
* impossibility for the patient to complete the forms
* impossibility to follow the patient
* patient with serious disease which impact the quality of life

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A prospective, non randomized, open, multicenter trial to evaluate non specific symptoms and quality of life (SF 36) before and after surgery for mild primary hyperparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2007-12; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
assessment of the evolution of neuropsychic disorders, digestive disorders, asthenia and polydipsia symptoms (non specific symptoms) one year after surgery for patients with moderate HPTI. | one year after surgery

SECONDARY OUTCOMES:
Evaluation of the quality of life with a quality of life questionnaire (SF36) given preoperatively and at months 3, 6, 12 | preoperatively and at months 3, 6, 12
evaluation of the evolution of neuropsychic disorders, digestive disorders, asthenia and polydipsia symptoms (non specific symptoms) at months 3 and 6 | at months 3 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Eric MIRALLIE, PU¨-PH, Principal Investigator — Nantes University Hospital
Locations (4):
- France (4):
  - Angers University Hospital, Angers
  - Limoges University Hospital, Limoges
  - Marseille University Hospital, Marseille
  - Nantes University Hospital, Nantes